CLINICAL TRIAL: NCT01976026
Title: Diversion of Flow in Intracranial VErtebral and Blood Blister-like Ruptured Aneurysms Trial Trial: A Randomized Trial Comparing Pipeline Flow Diversion and Best-Standard-Treatment
Brief Title: DIVERT: Diversion of Flow in Intracranial VErtebral and Blood Blister-like Ruptured Aneurysms Trial: A Randomized Trial Comparing Pipeline Flow Diversion and Best-Standard-Treatment
Acronym: DIVERT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Rare aneurysms. No patient enrolled at site.
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CE13.114
Record Dates: First submitted 2013-10-22; First posted 2013-11-05 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Ruptured Aneurysm of Intracranial Artery
Keywords: Flow Diversion; Aneurysm; Intracranial; Cerebral; Vertebral; blood blister-like; ruptured aneurysm; Pipeline Flow Diversion; Pipeline Flow Diverter; Best-Standard Treatment
MeSH Terms: conditions — Aneurysm; Aneurysm, Ruptured

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Endovascular treatment with flow diversion (Experimental): Endovascular treatment with flow diversion, including standard management of thrombo-embolic risk. The goal of the treatment procedure is (as usual) to prevent rebleeding, while keeping treatment-related risks as low as possible.
  This trial permits the interventionist or surgeon to use any device, technique or drug judged important to the safety and success of the endovascular or surgical procedure, at his/her discretion at any time during the procedure. It is imperative that the allocated procedure is conducted in the safest possible manner. The interventionist or surgeon may switch to an alternative BST or cross-over to the alternative treatment group, if it is in the best interest of the patient.
  Interventions: Device: Flow Diversion
- Best standard therapy (Active Comparator): May be any of the following:
  Conservative management when no surgical or endovascular treatment is considered possible or reasonable
  Conventional endovascular options including coiling with or without high-porosity stenting, and stent-in stent techniques
  Parent vessel occlusion, with or without bypass
  Surgical clipping or clip-wrapping (including parent vessel occlusion as a salvage procedure).
  Choice of best option is based on the location, anatomy, and particular circumstances, before randomization for this patient's aneurysm.
  This trial permits the interventionist or surgeon to use any device, technique or drug judged important to the safety and success of the endovascular or surgical procedure, at his/her discretion at any time during the procedure. The interventionist or surgeon may switch to an alternative BST or cross-over to the alternative treatment group, if it is in the best interest of the patient.
  Interventions: Device: Best Standard Therapy

INTERVENTIONS:
Device: Flow Diversion
  Arms: Endovascular treatment with flow diversion
Device: Best Standard Therapy
  Other Names: Best standard therapy, which may be any of the following:; B1. Conservative management when no surgical or endovascular treatment is considered possible or reasonable; B2. Conventional endovascular options including coiling with or without high-porosity stenting, and stent-in stent techniques; B3. Parent vessel occlusion, with or without bypass; B4. Surgical clipping or clip-wrapping (including parent vessel occlusion as a salvage procedure).
  Arms: Best standard therapy

SUMMARY:
The purpose of the DIVERT study is to provide a prudent, controlled clinical context for the use of flow diversion, a promising option of yet unproven benefit, in the care of patients with acute blood blister-like and dissecting intradural aneurysms. Hence DIVERT is a simple, multicenter, randomized trial integrated into daily practice. DIVERT addresses the clinical dilemma of whether the use of PED FD truly is a safe and effective alternative to best standard treatment, defined as conventional methods of treatment or in some cases, observation. Selection criteria are few, to facilitate the recruitment of most affected patients confronted with these difficult aneurysms that their physician judges suitable for PED FD. The trial does not obstruct clinical care, does not include extra tests or risks beyond what is necessary and proven beneficial. Endpoints are simple, clinical, meaningful, valuable and resistant to bias. Follow-up visits and tests are "routine', imposing no extra burden on clinical transactions. Data is collected in simple case-report forms filled by physicians.

DETAILED DESCRIPTION:
Ruptured blood blister-like (BB) and dissecting vertebral aneurysms are infrequent but devastating causes of subarachnoid hemorrhage (SAH), prone to acute rebleeding with poor clinical outcomes despite current surgical or endovascular treatment. Flow diversion (PED FD) with the Pipeline Endovascular Device (PED) is a promising treatment alternative to conventional management options.

The DIVERT trial is designed to provide a prudent, controlled clinical framework for offering the PED FD , a promising yet unproven option in the care of patients with acute blood blister-like or dissecting vertebral aneurysms. DIVERT is a care trial, designed as a simple, pragmatic, multicenter, randomized trial integrated into daily practice with inclusive selection criteria.

The investigators hypothesize that PED FD can decrease poor outcomes from 30 to 15%, compared to 'best standard treatment' (BST). BST is chosen prior to randomization amongst 4 options: observation, coiling with or without stenting, parent vessel occlusion or surgical clipping or wrapping. Patients are enrolled within 48 hours of SAH using standard 1:1 randomization between PED FD and BST after informed consent has been obtained from the patient or surrogate decision maker(s). Patients for whom no other option than PED FD appears feasible and safe will be included in a registry conducted alongside the trial.

Blister-like aneurysms and intradural dissections presenting with SAH have a high propensity for rebleeding and outcomes are poor in approximately one third of the cases, despite treatment using surgical or endovascular techniques.

ELIGIBILITY:
Inclusion Criteria:

* A patient affected with a blood blister-like aneurysm or a dissecting aneurysm, vertebral or at other sites, responsible for a recent subarachnoid hemorrhage (<14 days) for whom PED FD is considered an appropriate therapeutic option by the participating clinician. Current indications may be (but not restricted to) symptomatic blister-like aneurysms and dissecting intradural vertebral aneurysms.

Exclusion Criteria:

1. Severe allergy, intolerance or bleeding disorder that prohibit the use of Acetyl Salicylic Acid (ASA), clopidogrel or other platelet inhibitors
2. Acute hydrocephalus or intracranial hematomas necessitating urgent ventricular drainage or surgical evacuation (patients may be recruited after these urgent interventions have been performed)
3. Absolute contraindication to endovascular treatment or anesthesia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-11; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Neurological status of the patient | 3 months following treatment
  Neurological status graded according to the Rankin scale, defined as mRS>2, from any disease, treatment or other related causes.
Neurological status of the patient | at last follow-up (1 year following treatment, +/- 1 month)
  Neurological status graded according to the Rankin scale, defined as mRS>2, from any disease, treatment or other related causes.

SECONDARY OUTCOMES:
Modified Rankin Scale score | within a month following treatment, and at 3 and 12 months post-treatment
Successful PED FD deployment/aneurysm clip-ligation/aneurysm coiling, with patency of parent arteries | within 24 hours after procedure, if appropriate
Peri-operative complications | Within one month of treatment
  Peri-operative complications (ischemic strokes and intracranial hemorrhages), defined as any severe adverse effect.
Angiographic outcome | between 3-12 months following treatment
  Angiographic outcome (invasive or non-invasive imaging) (last observation carried forward)
Number of days of hospitalization | Within a month following procedure
Discharge disposition/location | within a month following procedure
  home; other hospital; rehabilitation facility; death
Any new stroke, neurological symptom or sign | during follow-up (between discharge and 1 year post-treatment)
Hospital re-admission | from initial discharge to one year following treatment
Hemorrhagic complications | within one year following treatment
  Hemorrhagic complications, in any body system, related to antiplatelet medication or not.
Re-treatment of the index aneurysm | Within one year following treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jean Raymond, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada